CLINICAL TRIAL: NCT01436981
Title: Observational Study on Papaverine During Cardiac Surgical Procedures
Brief Title: Pharmacokinetics of Pavaverine After Intraluminal Administration
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Klinikum Ludwigshafen (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head cardiovascular research, Johann Wolfgang Goethe University Hospital
Other Study IDs: PAV002-AHK
Record Dates: First submitted 2011-09-14; First posted 2011-09-20 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Injury of Internal Mammary Artery; Complications Due to Coronary Artery Bypass Graft
Keywords: papaverine; pharmacokinetic; CABG; Injury of Internal Mammary Artery; Complications Due to Coronary Artery Bypass Graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG with papaverine: Patients with CABG procedure
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — Preparation of artery mammaria interna
  Other Names: Paveron N

SUMMARY:
The purpose of this study is to determine the pharmacokinetic of papaverine after administration into the artery mammaria interna.

ELIGIBILITY:
Inclusion Criteria:

* CABG
* Administration of papaverine into mammaria interna

Exclusion Criteria:

* Allergy against papaverine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CABG patients
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of papaverine | 4 hours
  Serum probes will be analysed for the concentrations of papaverine.

CONTACTS AND LOCATIONS:
Overall Officials: Arndt H Kiessling, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Klinikum der Goethe Universität Frankfurt, Frankfurt am Main, Hesse, Germany